CLINICAL TRIAL: NCT06473675
Title: Hysterectomy With Adnexal Surgery Procedures With the DEXTER Robotic System
Brief Title: Hysterectomy With Adnexal Surgery Procedures With the DEXTER Robotic System (The HYPER Study)
Status: Completed | Type: Observational
Sponsor: Distalmotion SA (Industry)
Collaborators: Confinis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-01
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hysterectomy
MeSH Terms: interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Hysterectomy with adnexal surgery — Robotic-assisted and laparoscopic hysterectomy with adnexal surgery for benign disease.

SUMMARY:
This study aims to confirm the perioperative and early postoperative safety and clinical performance (efficacy) of the Dexter Robotic System, in patients undergoing robotic-assisted and laparoscopic hysterectomy with adnexal surgery for benign disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Patients planned to undergo elective robot-assisted and laparoscopic hysterectomy with adnexal surgery for benign disease; using one camera port, two ports for the manipulating instruments, and additional ports as needed.

Exclusion Criteria:

* Morbidly obese patients (BMI > 40)
* Any relative and absolute contraindications for the use of conventional endoscopes and endoscopic surgical instruments
* Need for robotic stapling, advanced energy delivery, ultrasound, cryoablation and microwave energy delivery
* Bleeding diathesis
* Pregnancy
* Patients with pacemakers or internal defibrillators
* Any planned concomitant procedures
* Patient deprived of liberty by administrative or judicial decision.
* Participation in another interventional clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing a hysterectomy with adnexal surgery for benign disease.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
primary safety endpoint | up to 42 days
  occurrence of Clavien - Dindo grades III-V adverse events
primary performance endpoint | intraoperative
  successful completion of the Dexter-assisted procedure, i.e. free of any conversion to an open or fully laparoscopic surgical approach

CONTACTS AND LOCATIONS:
Locations (4):
- Groupe Hospitalier Saintes - Saint-Jean-d'Angély, Saintes, France
- Switzerland (3):
  - Kantonsspital Baden, Baden
  - Inselspital Bern, Bern
  - Spitäler FMI AG, Interlaken

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gulz M, Bodet ML, Streich M, Habegger A, Heubner M, Erhardt D, Bogdanovic B, Mueller MD. Multicenter evaluation of the DEXTER(R) Robotic Surgery System for Total Hysterectomy with Adnexal Surgery. J Robot Surg. 2025 Sep 26;19(1):634. doi: 10.1007/s11701-025-02647-0. PMID 40999110